CLINICAL TRIAL: NCT00238849
Title: Phase II Study of Oxaliplatin in Combination With Navelbine for the Second-Line Treatment of Advanced and Metastatic Non-Small Cell Lung Cancer
Brief Title: Phase II Study of Oxaliplatin and Navelbine for Second-Line Treatment of Advanced NSCLC.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Integrated Community Oncology Network (Other)
Collaborators: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OX-03-087; ELVIS II
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2005-10-14 (Estimated); Status verified 2005-10

CONDITIONS: Previously Treated Metastatic Non-Small Cell Lung Cancer
Keywords: Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin

SUMMARY:
The purpose of this study is to determine the response rate to treatment with oxaliplatin and Navelbine in patients with previously treated NSCLC. Oxaliplatin and Navelbine have not been clinically evaluated yet. However, Navelbine has been safely administered with other platinum compounds.

DETAILED DESCRIPTION:
This is a non-randomized trial for patients with previously treated Non-small cell lung cancer. Each patient will receive 6 cycles of chemotherapy consisting of Oxaliplatin and Navelbine. Oxaliplatin is given intravenously every 21 days and Navelbine is administered Intravenously on day 1 and day 8 every 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic non-small cell lung cancer that has recurred, progressed, or failed to respond to previous systemic chemo.
* Measurable disease
* Good performance status (ECOG 0,1 or 2)

Exclusion Criteria:

* Previously treated with Oxaliplatin or Navelbine
* Symptomatic CNS metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40

PRIMARY OUTCOMES:
Efficacy

SECONDARY OUTCOMES:
Time to progression
Duration of response
Survival
Toxicity profile

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Marsland, MD, Principal Investigator — Integrated Community Oncology Network
Locations (2):
- United States (2):
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Integrated Community Oncology Network, Orange Park, Florida